CLINICAL TRIAL: NCT03939468
Title: A HYbrid APproach Evaluating A DRug-Coated Balloon in Combination With A New Generation Drug-Eluting Stent in the Treatment of De Novo Diffuse Coronary Artery Disease
Brief Title: Drug-Coated Balloon in Combination With New Generation Drug-Eluting Stent for de Novo Diffuse Disease Treatment
Acronym: HYPER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, ALFONSO IELASI, Principal Investigator, I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Other Study IDs: HYPER v3
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug Coated Balloons; Drug Eluting Stent; Diffuse Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Cohort: Patient with diffuse CAD disease treated with hybrid strategy (DES+DCB)
  Interventions: Device: DES+DCB

INTERVENTIONS:
Device: DES+DCB — A hybrid strategy is defined as overlapping or slightly (2-3 mm) superimposing a new generation DES implantation for a de novo lesion (located in the larger, more proximal part of the vessel) and DCB inflation for a concomitant de novo small vessel disease

SUMMARY:
A Pilot Observational Study to evaluate safety and efficacy of the hybrid approach DES/DCB in treating de-novo diffuse lesions

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-arm, multi-center, pilot, noninterventional study whose aim is to assess the feasibility and the clinical outcomes of using the Restore DCB (Cardionovum GmbH, Bonn, Germany) in combination ("hybrid approach") with a new generation DES (type at operator's discretion) for the treatment of diffuse CAD encountered in daily clinical practice. The rationale of the proposed strategy derives from the characteristics of DCB in treating the atherosclerotic disease without leaving a permanent structure in the vessel especially in case of diffuse CAD -avoiding a long metallic, permanent cage within extended coronary segments

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with stable or unstable CAD eligible for PCI (according to the international guidelines) because of diffuse CAD involving segments suitable for a hybrid approach;
* Signed Patient Informed Consent/Data Release Form

Exclusion Criteria:

1. Age <18 years;
2. Cardiogenic shock;
3. Pregnancy or breastfeeding;
4. Infarct-artery max diameter (within planned device deployment segment) <2.0 or >5.0 mm;
5. Comorbidities with life expectancy <6 months;
6. Severe calcification or/tortuosity proximally or at the DCB target segment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable or unstable CAD eligible for PCI (according to International guidelines) due to diffuse disease (located in the same vessel) suitable for a "hybrid approach" (see below) will be enrolled after signing the informed consent. A hybrid strategy was defined as overlapping or slightly (2-3 mm) superimposing a new generation DES implantation for a de novo lesion (located in the larger, more proximal part of the vessel) and DCB inflation for a concomitant de novo small vessel disease (located in the smaller distal segment or at a side branch of a bifurcation in the same coronary artery). Diffuse disease is defined as CAD≥28 mm in length involving distal segments or side branches of a bifurcation lesion with a reference vessel diameter (RVD) considered suitable for a hybrid approach in case of ≥2.75 mm RVD for a DEStarget segment and ≥2.0 mm to <2.75 mm RVD for a DCB-target segment.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
DOCE at 12 Months | 12 Months
  A device oriented composite end-point (DOCE) of cardiac death, target vessel myocardial infarction (TV-MI) and ischemia-driven target lesion revascularization (ID-TLR) in the DES- and/or the DCB-treated segment within 12 months after the index procedure

SECONDARY OUTCOMES:
Procedural Success | At procedure
  Procedural success defined as both DCB/DES delivery and implantation at the "target" lesion site with <30% diameter stenosis (DS) in the DCB-treated segment and <10% DS in the DES-treated segment and distal TIMI 3 flow.
Peri-procedural myocardial infarction | Pre-discharge
  Peri-procedural myocardial infarction defined as an elevation of cardiac biomarkers (troponin or creatine kinase-myocardial band) >3 times the upper limit of normal
DOCE | Pre-discharge, 30 days, 6 months, 12 months
  DOCE and its singular components (cardiac death, any TV-MI excluding peri-procedural MI, ID-TLR ) in-hospital, (within 7 days after PCI) and at 30-day, 6-month, 1-year follow-up
Thrombosis | 12 months
  Any definite/probable DES- or DCB-treated segment thrombosis (in-hospital, within 7 days after PCI and at 30-day, 6month, 1-year follow-up).
Flow-limiting dissection | 12 months
  Flow-limiting dissection (type C-F waiting 3 minutes after DCB inflation) requiring additional DES implantation in the DCB-treated segment

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Presidio Ospedaliero di Rho, Rho, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Istituto Clinico S.Anna, Brescia
  - ASST Ospedale Cremona, Cremona
  - Istituto Clinico S.Ambrogio, Milan
  - Policlinico Casilino, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Costopoulos C, Latib A, Naganuma T, Sticchi A, Figini F, Basavarajaiah S, Carlino M, Chieffo A, Montorfano M, Naim C, Kawaguchi M, Giannini F, Colombo A. The role of drug-eluting balloons alone or in combination with drug-eluting stents in the treatment of de novo diffuse coronary disease. JACC Cardiovasc Interv. 2013 Nov;6(11):1153-9. doi: 10.1016/j.jcin.2013.07.005. PMID 24262615
- [Background] Ielasi A, Miyazaki T, Geraci S, Testa L, Abdel-Wahab M, Kawamoto H, Ruparelia N, Sato T, Caramanno G, Bedogni F, Tespili M, Colombo A, Latib A. Hybrid strategy with a bioresorbable scaffold and a drug-coated balloon for diffuse coronary artery disease: the "no more metallic cages" multicentre pilot experience. EuroIntervention. 2016 Apr 8;11(14):e1589-95. doi: 10.4244/EIJV11I14A309. PMID 27056119
- [Background] Tang Y, Qiao S, Su X, Chen Y, Jin Z, Chen H, Xu B, Kong X, Pang W, Liu Y, Yu Z, Li X, Li H, Zhao Y, Wang Y, Li W, Tian J, Guan C, Xu B, Gao R; RESTORE SVD China Investigators. Drug-Coated Balloon Versus Drug-Eluting Stent for Small-Vessel Disease: The RESTORE SVD China Randomized Trial. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2381-2392. doi: 10.1016/j.jcin.2018.09.009. PMID 30522667
- [Background] Ielasi A, Buono A, Pellicano M, Tedeschi D, Loffi M, Donahue M, Regazzoli D, De Angelis G, Danzi G, Reimers B, Tespili M. A HYbrid APproach Evaluating a DRug-Coated Balloon in Combination With a New-Generation Drug-Eluting Stent in the Treatment of De Novo Diffuse Coronary Artery Disease: The HYPER Pilot Study. Cardiovasc Revasc Med. 2021 Jul;28:14-19. doi: 10.1016/j.carrev.2020.07.036. Epub 2020 Jul 31. PMID 32933874
- [Derived] Buono A, Pellicano M, Regazzoli D, Donahue M, Tedeschi D, Loffi M, Zimbardo G, Reimers B, Danzi G, DE Blasio G, Tespili M, Ielasi A. Procedural and one-year outcomes following drug-eluting stent and drug-coated balloon combination for the treatment of de novo diffuse coronary artery disease: the HYPER Study. Minerva Cardiol Angiol. 2024 Apr;72(2):163-171. doi: 10.23736/S2724-5683.23.06352-4. Epub 2023 Sep 13. PMID 37705369